CLINICAL TRIAL: NCT04739618
Title: A Phase 2 Trial of Non-ablative Cryosurgical Freezing and Multiplex Immunotherapy in Patients With Metastatic Solid Cancer
Brief Title: Metastatic Solid Cancer Clinical Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunSYS, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEDROCK 1001
Record Dates: First submitted 2021-01-14; First posted 2021-02-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab; Ipilimumab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: Male or female subjects greater than 18 years of age with histologically-proven metastatic cancer with at least one imaging- or histologically- proven metastases to lymph nodes, bone, or soft tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm. Subjects receiving treatment. (Experimental): Efficacy of Non-ablative Cryosurgical Freezing and Multiplex Immunotherapy as determined by overall response rate of radiographic changes according to iRECIST criteria
  Interventions: Drug: Keytruda Injectable Product; Drug: Yervoy Injectable Product; Drug: GM-CSF; Procedure: Non-ablative Cryosurgical freezing

INTERVENTIONS:
Drug: Keytruda Injectable Product — PD-1 inhibitor antibody
  Other Names: pembrolizumab
Drug: Yervoy Injectable Product — Anti-CTLA-4 antibody
  Other Names: ipilimumab
Drug: GM-CSF — 1 mL injected into each non-ablative cryosurgical freezing zone. Daily injection administered subcutaneously. 250 mcg daily injections for a total of 25 days after each treatment.
  Other Names: sargramostim
Procedure: Non-ablative Cryosurgical freezing — To induce immediate necrosis and necroptosis and a rim of injured cancer cells, thereby exposing a complete range of patient-specific tumor antigens that are specific to the treated subject.

SUMMARY:
This study seeks to estimate the potential efficacy of the study treatment, as well as the occurrence of adverse events.

DETAILED DESCRIPTION:
Non-ablative Cryosurgical Freezing (limited to 1.5 cm diameter single freeze within the cancer (up to two cancer sites selected and treated)) will release intact antigens to prime the immune system. The study treatment immunotherapeutic drugs (PD-1 inhibitor monoclonal antibody Keytruda (pembrolizumab), anti-CTLA-4 monoclonal antibody ipilimumab, and GM-CSF) will then be sequentially injected directly into each of the treated cancer sites immediately following Non-ablative Cryosurgical Freezing. Daily subcutaneous GM-CSF injections will also be administered subsequently. It is speculated that neoantigens released from the cryo-frozen necrotic cancer will be available in the vicinity of the Non-ablative Cryosurgical Freezing field immediately following the procedure. Immature dendritic cells attracted to the injection site will internalize neoantigens to become activated to recognize cancer-specific antigenic proteins. The activated dendritic cells will recruit killer T-cells to the injection site to attack cancer cells, and then migrate through the lymphatic system to sites of metastases, targeting cancer-specific neoantigens and recruiting more killer T-lymphocytes to destroy other cancer cells harboring the precise antigenic epitopes (abscopal (bystander) effect). In this way, dendritic cells are capable of initiating cell-mediated systemic immune response in combination with cytotoxic killer T-cells. Regulatory T lymphocytes, which have been implicated in dampening or halting cell-mediated, antigen-specific immune responses, will be selectively depleted by anti-CTLA-4 monoclonal antibodies, intra-tumoral GM-CSF, and GM-CSF. Intra-tumoral injection of the immunotherapeutic medications assists in stimulating and harnessing the local and systemic immune response. GM-CSF prolongs the immune response. Using this combination of therapies, referred to as YourVaccxTM, it is thought that a clinically significant systemic anti-cancer immune response might be elicited. Intra-tumoral injection of drugs will likely offer fewer side effects than systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Have a performance status of 0-2 on the ECOG Performance Scale.
* Have a life expectancy of 6 months or more as determined by treating physician.
* Have exhausted all other standard therapies; Have failed available therapy or are not a candidate for, or refuse available therapy (i.e. concerned with high adverse events rate in available therapy or outcome worse than disease); or failure of prior chemotherapy.
* Histologically-documented solid cancer. All subjects must submit their primary tumor or metastatic pathology specimens and laboratory and imaging reports to ImmunSYS where they will be centrally reviewed. Central ImmunSYS pathologic review is not required for screening but rather for confirmation of diagnosis and histologic subtype of cancer. Local pathologic review is sufficient for eligibility determination.
* Measurable disease as defined using iRECIST criteria and identified by radiographic imaging (Imaging should be current within the past three months of subject entering the study; if not repeat imaging must be done prior to enrollment.). In order to be eligible, the patient must have at least one metastatic bone and/or metastatic soft tissue site, lymph node site, and/or bone site with cancer mass measuring 1.5 cm or more in diameter based on soft tissue, lymph node, and/or bone lesions as defined by any of the following:

  * Any soft tissue lesion defined by imaging deemed by the physician to be consistent with distant metastatic disease. For patients undergoing PSMA PET (prostate cancer patients only), only PSMA avid lesions that have a CT or MRI correlate consistent with metastasis will be counted as a site of metastasis.
  * Metastatic lymph node disease defined by imaging. Any lymph node ≥1 cm in shortest dimension will be noted as involved with disease.
  * Bone metastases defined by bone imaging. If the patient has technetium bone scan and/or NaF PET performed, either study may be used for documenting metastases; both scans do not need to show the number of metastases required for study entry. For patients undergoing PSMA PET (prostate cancer patients only), only PSMA-avid lesions that are consistent with metastasis will be counted as a site of metastasis.
* The effects of the medications in this protocol on the developing human fetus are unknown. Any subject treated or enrolled on this protocol must agree to use adequate contraception prior to the first dose of study therapy, for the duration of the study participation, and for 120 days after the last dose of study therapy.
* Their partners will also be encouraged to use proper method of contraception.
* Acceptable initial laboratory values within 14 days of treatment initiation according to the following:

ANC ≥ 1500/µl Hemoglobin ≥ 9.0 g/dL(prior transfusion permitted) Platelet count ≥ 100,000/µl Creatinine ≤ 2.0 x the institutional upper limit of normal (ULN) OR creatinine clearance >30 ml/min Potassium ≥ 3.5 mmol/L (within institutional normal range) Bilirubin ≤ 1.5 x ULN (unless documented Gilbert's disease) SGOT (AST) ≤ 2.5x ULN, or <5x ULN in patients with documented liver metastases SGPT (ALT) ≤ 2.5x ULN or <5x ULN in patients with documented liver metastases Albumin >2.5 mg/dL Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

Deviation from these values is allowed at the discretion of the treating investigator.

* NOTE: Women of child-bearing potential will be tested for pregnancy (which must be negative) before treatment is given. Acceptable range is < 5 mIU/mL
* No active major medical or psychological problems that could be complicated by study participation.

Exclusion Criteria:

* Is currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has bone metastasis as the only site of disease.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment, with the exception of steroids for adrenal insufficiency in which case prednisone <10mg/day or its equivalent is allowed.
* Has a performance status of 3-5 on the ECOG Performance Scale.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to monoclonal antibodies such as Keytruda (pembrolizumab) or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Is taking any current medication known to interfere with serum PSA concentration or radiographic extent of cancer (e.g., Enzalutamide, hormonal therapy) within 30 days for non-depot or 90 days for depot of start of treatment.
* Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Persisting toxicity related to prior therapy (NCI CTCAE v.5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, Grade 2 anemia, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include carcinoid, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs), including but not limited to systemic or cutaneous lupus erythematosus, cutaneous psoriasis, psoriatic arthritis, rheumatoid arthritis, scleroderma, sicca syndrome, polymyalgia rheumatica, polyarteritis nodosa, granulomatous polyangiitis, microscopic polyangiitis, polyarteritis nodosa, temporal arteritis, giant-cell arteritis, dermatomyositis, Kawasaki disease. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, hydroxychloroquine, etc.) is not considered a form of systemic treatment.
* Has known recent (within 2 years) history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorder or any other condition that would interfere with cooperation with the requirements of the trial in the opinion of the Physician-investigator.
* Pregnant and/or expecting to bear or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 30 days.
* Personal representative (family member or friend) withholds consent for any reason.
* Unable for any reason to understand the consent form and other written information and freely give written informed consent.
* Score less than 12.0 (out of possible maximum of 20) on the UBACC Capacity to Consent Assessment Instrument.
* Hypersensitivity to GM-CSF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Non-ablative Cryosurgical Freezing and Multiplex Immunotherapy as determined by overall response rate of radiographic changes according to iRECIST criteria. | baseline to 8 weeks after end of treatment (approximately 5 months)
  Efficacy of Non-ablative Cryosurgical Freezing and Multiplex Immunotherapy as determined by overall response rate of radiographic changes according to iRECIST criteria.

SECONDARY OUTCOMES:
Efficacy of Non-ablative Cryosurgical Freezing and Multiplex Immunotherapy as determined by RECIST1.1 criteria | baseline to 8 weeks after end of treatment (approximately 5 months)
  Overall response rate as determined using RECIST1.1 radiographic response

OTHER OUTCOMES:
Radiographic progression-free survival (rPFS) | baseline to 8 weeks after end of treatment (approximately 5 months)
  rPFS as determined with both RECISTS1.1 and iRECIST criteria
Best overall response of confirmed PR or CR by independent radiology review | baseline to 8 weeks after end of treatment (approximately 5 months)
  Best overall response of confirmed PR or CR by independent radiology review
Time to progression (TTP) based on independent radiology review | baseline up to 8 weeks after last treatment
  Time to cancer progression is measured from the date of first study treatment until the date of cancer progression.
Overall survival | 3 years
  Number and percent of participants that are alive.
Incidence of AEs/SAEs | baseline to 8 weeks after the last treatment
  An AE is any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity. Incidence was defined as the number of participants who experienced an adverse event within their period of participation in this study. Incidence of adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Severity of AEs/SAEs | baseline through 8 weeks after the last treatment
  Severity of AEs/SAEs
Duration of AEs/SAEs | baseline through 8 weeks after the last treatment
  Duration of AEs/SAEs
The time to objective disease progression | baseline through 8 weeks after the last treatment (Safety Follow-Up)
  Data will be collected for the design of future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Onik, M.D., Principal Investigator — ImmunSYS, LLC
Locations (2):
- United States (2):
  - Vincere Cancer Center, Scottsdale, Arizona
  - Florida Endovascular and Interventional, Miami Lakes, Florida